CLINICAL TRIAL: NCT04457232
Title: PET Biodistribution Study of 68Ga-FAPI-46 in Patients With Prostate Cancer: A Prospective Exploratory Biodistribution Study With Histopathology Validation
Brief Title: Prospective Exploratory Study of FAPi PET/CT in Prostate Cancer With Histopathology Validation
Acronym: FAPI PET Prost
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-000177; NCI-2020-02712 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-000177 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Malignant Neoplasm in the Prostate Gland; Prostate Carcinoma; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — FAPI-46; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Basic Science (68Ga-FAPi-46 PET/CT) (Experimental): Patients receive 68Ga-FAPi-46 IV and undergo PET/CT imaging over 20-50 minutes.
  Interventions: Procedure: Computed Tomography; Other: Gallium Ga 68 FAPi-46; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT imaging
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Gallium Ga 68 FAPi-46 — Given IV
  Other Names: 68Ga-FAPi-46; Gallium-68-FAPi-46
Procedure: Positron Emission Tomography — Undergo PET/CT imaging
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This exploratory study investigates how a new imaging technique called FAPI PET/CT can determine where and to which degree the FAPI tracer (68Ga-FAPi-46) accumulates in normal and cancer tissues in patients with prostate cancer. Because some cancers take up 68Ga-FAPi-46 it can be seen with PET. FAP stands for Fibroblast Activation Protein. FAP is produced by cells that surround tumors. The function of FAP is not well understood but imaging studies have shown that FAP can be detected with FAPI PET/CT. Imaging FAP with FAPI PET/CT may in the future provide additional information about various cancers including prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the biodistribution of gallium 68Ga-FAPi-46 in normal and cancer tissues of patients with prostate cancer.

SECONDARY OBJECTIVES:

I. To evaluate whether 68Ga-FAPi-46 and gallium Ga 68-labeled PSMA-11 (68Ga-PSMA-11) accumulation observed by positron emission tomography (PET) correlates with the amount of fibroblast activation protein (FAP) and prostate specific membrane antigen (PSMA) in excised cancer tissue, respectively.

II. To assess the 68Ga-FAPI-46 biodistribution correlation with 68Ga-PSMA-11.

OUTLINE:

Patients receive 68Ga-FAPi-46 intravenously (IV) and undergo PET/computed tomography (CT) imaging over 20-50 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a 68Ga-PSMA-11 PET/CT scan within 3 months of enrollment
* Patients who are scheduled to undergo surgical excision or biopsy of a prostate cancer primary, recurrent or metastatic lesion
* Patients can provide written informed consent
* Patients are able to remain still for duration of imaging procedure (up to one hour)

Exclusion Criteria:

* Patients with any new prostate therapy between the PSMA PET/CT and the FAP inhibitor (FAPI) PET/CT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
To define and document the biodistribution of gallium 68Ga-FAPi-46 in normal and cancer tissues of patients with prostate cancer | 60 minutes after tracer injection
  To quantify tumor tissue and normal background organs positron emission tomography (PET) tracer uptake by semi-quantitative analysis (unit/metrics = standardized uptake values [SUV], SUVmean and SUVmax.

SECONDARY OUTCOMES:
To evaluate whether 68Ga-FAPi-46 accumulation observed by PET correlates with the amount of fibroblast activation protein (FAP) assessed by immunohistochemistry (IHC) in excised cancer tissue | Up to date of surgery (range 1-60 days)
  68Ga-FAPi-46 tumor SUVs will be correlated with FAP expression from surgically resected tumors. IHC will be scored with a semi-quantitative scoring system that accounts for staining intensity (0-2, where 0 is negative, 1 is weak, 2 is strong and eq. stands for equivocal). Correlations will be sought using least square regression analysis.
To assess the 68Ga-FAPI-46 biodistribution correlation with 68Ga-PSMA-11 PET imaging | 60 minutes after tracer injection
  The 68Ga-PSMA-11 and 68Ga-FAPI-46 tracer biodistribution will be described by mean and maximum standardized uptake values (SUVmean and SUVmax) and tested for correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States